CLINICAL TRIAL: NCT02428153
Title: Investigation Of Muscle-Tendon Unit By Ultrasound After Static And Dynamic Stretching
Brief Title: Effect Of Static And Dynamic Stretching On Muscle Tendon Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Funda DEMIRTURK, Assoc. Prof., Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15-KAEK-025 (Ethics Committee)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: static stretching; dynamic stretching; muscle-tendon unit; ultrasound; Subjects
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cases (Experimental): static and dynamic stretching exercises
  Interventions: Other: stretching exercises

INTERVENTIONS:
Other: stretching exercises — static stretching exercise of 5 repetitions, with a duration of 45 seconds to the right gastrocnemius muscle and dynamic stretching exercise of 5 repetitions, with a duration of 45 seconds to the cases' left gastrocnemius muscles
  Other Names: static stretching exercise; dynamic stretching exercise

SUMMARY:
The purpose of this study is to investigate the acute effects of two different types of muscle stretching (static and dynamic) on muscle-tendon unit of gastrocnemius muscle by ultrasound and to follow how long the stretching effects are sustained.

DETAILED DESCRIPTION:
Muscle stretching is a very common practice applied in warm-up process in order to enhance performance in sports and to prevent or decrease the risk of sports injury. Muscle stretching is also used for therapeutic purposes in many clinical conditions.

It is generally performed in either static or dynamic manner. Muscle is brought to its lengthened position and is held at that point for a certain period of time in static stretching (SS). In dynamic stretching (DS), however, active movements of muscle take the joint through the range of motion and creates a stretch, but the muscle is not held in the end position.

Although recent studies suggest that static stretching has adverse effects on performance, reduces maximal muscle force and is not successful in preventing non-contact injuries, as believed so; and the dynamic type therefore gaining popularity; it is reported that flexibility and range of motion can be improved by stretching as a consequence of the decrement in muscle stiffness. However, the effects of stretching depend on the type, duration and timing of stretching and there is still debate over which prescription provides the best results in terms of flexibility, power, performance or injury protection. And what happens to the viscoelastic properties of a muscle when it is stretched statically or dynamically is still not well documented. Ultrasound seems to be a good option as it offers an objective and a non-invasive way to expose the alteration in muscles and tendons due to stretching.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males,
* aged between 18-30 years

Exclusion Criteria:

* Cases with history of recent musculoskeletal injuries or neurological diseases.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
muscle-tendon unit length | before stretching exercises and just after the stretching exercises and 5, 15 and 30 minutes after stretching
  change in muscle tendon unit property with static and dynamic exercises will be followed by ultrasound before, right after and 5, 15 and 30 minutes after the stretching exercises
pennation angle | before stretching exercises and just after the stretching exercises and 5, 15 and 30 minutes after stretching
  change in pennation angle of the gastrocnemius muscle with static and dynamic exercises will be followed by ultrasound before, right after and 5, 15 and 30 minutes after the stretching exercises
muscle thickness | before stretching exercises and just after the stretching exercises and 5, 15 and 30 minutes after stretching
  change in muscle thickness of the gastrocnemius muscle with static and dynamic exercises will be followed by ultrasound before, right after and 5, 15 and 30 minutes after the stretching exercises

SECONDARY OUTCOMES:
range of ankle dorsiflexion | before stretching exercises and just after the stretching exercises and 5, 15 and 30 minutes after stretching
  change in range of ankle dorsiflexion with static and dynamic exercises will be followed by ultrasound before, right after and 5, 15 and 30 minutes after the stretching exercises

CONTACTS AND LOCATIONS:
Overall Officials: Funda DEMIRTURK, PhD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)